CLINICAL TRIAL: NCT00560703
Title: Efficacy and Safety of COL-101 for the Treatment of Blepharitis in Patients With Facial Rosacea
Brief Title: Treatment of Patients With Blepharitis and Facial Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COL-101-BLEPH-201
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-12

CONDITIONS: Blepharitis; Meibomianitis; Dry Eye
MeSH Terms: conditions — Blepharitis; Meibomitis; Dry Eye Syndromes | interventions — Doxycycline; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- COL-101 (doxycycline, USP) capsules (Active Comparator): COL-101
  Interventions: Drug: COL-101 (doxycycline, USP) capsules
- Placebo (Placebo Comparator): Sugar capsule
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: COL-101 (doxycycline, USP) capsules — 40mg, once per day for 84 days
  Arms: COL-101 (doxycycline, USP) capsules
Drug: placebo — sugar capsule
  Arms: Placebo

SUMMARY:
To determine the safety and efficacy of sub-antimicrobial dose COL-101 in the treatment of patients who have both blepharitis and facial rosacea

ELIGIBILITY:
Inclusion Criteria:

* blepharitis
* facial rosacea

Exclusion Criteria:

* pregnant or nursing women
* allergy to tetracyclines
* recent eye surgery
* past or current use of isotretinoin
* patients who are achlorhydric
* patients who have had gastric by-pass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (8):
- United States (8):
  - Pleasant Valley Ophthalmology, Little Rock, Arkansas
  - Warren Scherer, MD, Naples, Florida
  - Kentucky Lions Eye Center, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - Marguerite McDonald, MD, Lynbrook, New York
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Anita Nevyas-Wallace, MD, Bala-Cynwyd, Pennsylvania
  - Tanner Clinic, Layton, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment time was approximately 6 months in 8 US clinics.
Pre-assignment Details: Subjects were screened for eligibility within 6 weeks prior to the baseline visit. This 12-week study employed a two-treatment, parallel-group design with subjects randomized in a 2:1 ratio to active drug or placebo.
Groups:
- COL-101 (Doxycycline, USP) Capsules: 40 MG, Once per day for 84 days
- Placebo: Sugar capsule, once per day for 84 days
Period: Overall Study
Arm/Group | COL-101 (Doxycycline, USP) Capsules | Placebo
Started | 46 | 24
Completed | 46 | 18
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COL-101 (Doxycycline, USP) Capsules | Placebo | Total
Number analyzed (Participants) | 46 | 24 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 15 | 51
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (13.46) | 58.2 (14.27) | 55.7 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 13 | 43
  Male | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 46 | 24 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Bulbar Conjunctival Hyperemia
Description: Bulbar conjunctival hyperemia will be assessed using an ordered categorical value ranging from 0 (Clear) to 4 (Severe). Hyperemia is graded on the following scale and half scores are acceptable:
  None (0) = normal Mild (1) = slight localized injection Moderate (2) = pink color Severe (3) = red color Very Severe (4) = marked dark redness
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COL-101 (Doxycycline, USP) Capsules | Placebo
Number analyzed (Participants) | 46 | 24
Scores on a scale | -0.61 (0.797) | -0.60 (0.707)
Statistical Analysis 1: Comparison: COL-101 (Doxycycline, USP) Capsules vs Placebo; Test type: Non-Inferiority or Equivalence — Power calculation for this endpoint was driven by the assumptions made for the OSDI analysis; p = 0.578, ANCOVA

2. Primary Outcome: Change in Ocular Surface Disease Index (OSDI)
Description: OSDI is calculated based following formula using 12-question Ocular Surface Disease questionnaire (with each question scored 0-4):
  OSDI = (D/E)x25, where D = Sum of all scores for questions answered E = Total number of questions answered (not including questions answered NA)
  Range of OSDI is 0 to 100 (higher score indicates worse condition).
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | COL-101 (Doxycycline, USP) Capsules | Placebo
Number analyzed (Participants) | 46 | 24
Scores on a scale | -5.15 (14.002) | -8.70 (17.719)
Statistical Analysis 1: Comparison: COL-101 (Doxycycline, USP) Capsules vs Placebo; It was anticipated that the difference between the treatment groups in mean reduction from baseline in OSDI scores will be approximately 7 points. A pooled standard deviation of 9.0 for the mean change from baseline OSDI score is expected. Under those assumptions a total of approximately 63 evaluable patients (42 COL-101 patients and 21 placebo patients) is sufficient to provide 80% power. The planned enrolment should provide enough evaluable patients to meet these assumptions; Test type: Superiority or Other; p = 0.293, ANCOVA

ADVERSE EVENTS:
Arm/Group | COL-101 (Doxycycline, USP) Capsules | Placebo
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/24
Other Adverse Events (participants affected / at risk) | 5/46 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COL-101 (Doxycycline, USP) Capsules (N=46) | Placebo (N=24)
Migraine headache (Nervous system disorders) | 1 (1) | 0 (0)
non-hodgkin's lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COL-101 (Doxycycline, USP) Capsules (N=46) | Placebo (N=24)
headache (Nervous system disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No